CLINICAL TRIAL: NCT02384876
Title: Determination of the Optimal Dose of Ephedrine in Intraoperative Arterial Hypotension of Newborns and Infants up to 6 Months of Age. A Randomized, Controlled, Open-label, Dose Escalation Study.
Brief Title: Determination of the Optimal Dose of Ephedrine in Intraoperative Arterial Hypotension of Newborns and Infants up to 6 Months of Age.
Acronym: EPHEDRINE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL14_0248; 2014-004190-16 (EudraCT Number)
Record Dates: First submitted 2015-02-27; First posted 2015-03-10 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Intraoperative Arterial Hypotension; Infant, Newborn
Keywords: pediatric; intraoperative arterial hypotension; ephedrine; general anesthesia
MeSH Terms: interventions — Ephedrine; Organization and Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ephedrine, dose : 0.6, 0.8, 1.0, 1.2 and 1.4 mg/kG (Experimental): Dose escalation: 6 successive cohorts with a maximal increasing dose
  Interventions: Drug: Ephedrine 30mg/10mL injectable solution, single administration, dose : 0.6, 0.8, 1.0, 1.2 and 1.4 mg/kG
- Ephedrine, dose : 0.1 mg/kG, reference dose (Active Comparator): Reference dose
  Interventions: Drug: Ephedrine 30mg/10mL injectable solution, single administration, dose : 0.1 mg/kG.

INTERVENTIONS:
Drug: Ephedrine 30mg/10mL injectable solution, single administration, dose : 0.6, 0.8, 1.0, 1.2 and 1.4 mg/kG
  Arms: Ephedrine, dose : 0.6, 0.8, 1.0, 1.2 and 1.4 mg/kG
Drug: Ephedrine 30mg/10mL injectable solution, single administration, dose : 0.1 mg/kG.
  Arms: Ephedrine, dose : 0.1 mg/kG, reference dose

SUMMARY:
The incidence of arterial hypotension under general anesthesia using sevoflurane is particularly high in newborns and infants up to 6 months of age. A decrease of 20% of the initial mean blood pressure (mBP) is the definition of significant arterial hypotension in adults and children. In adults, intraoperative arterial hypotension is associated with an increase of intraoperative mortality and a certain neurological morbidity. In infants under 6 months of age, neurological disorders have been reported following general anesthesia. Neurotoxicity of hypnotics is often incriminated as should be the episodes of arterial hypotension.

Current management of hypotension uses vascular filling with crystalloids and vasopressive amines in second intention. Dopamine is the most frequently used amine. Ephedrine can also be used. Ephedrine is particularly interesting because of its action on both α and β receptors and its mode of administration: one dose and peripheral access.

Only one study is available in children from birth to adulthood; it demonstrates a lower hemodynamic response in infants than in adults, when administered a low dose of Ephedrine (0.1 to 0.2 mg/kg). A recent retrospective cohort suggests an under efficacy of low doses and the use of higher doses than those recommended.

The primary objective is to determine the optimal dose of ephedrine (dose of ephedrine associated with a difference of proportion of newborns/infants in therapeutic success of 55%) compare to the reference dose of 0.1mg/kg as a first line treatment of intraoperative arterial hypotension.

Secondary objectives:

* Return to a mBP superior to 38mmHg post Ephedrine administration.
* To assess occurrence of hypoxemic events during anesthesia.
* To assess tolerance of ephedrine. One hundred and twenty newborn and infants up to 6 months of age will be recruited in 3 sites of the Rhone Alpes Auvergne area over 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Newborns or infants < 6 months of age,
* boys and girls,
* premature or not,
* requiring general anesthesia induced by sevoflurane
* who presents during anesthesia a decrease of blood pressure superior to 20% of the basal mBP (measured prior to surgery) despite of vascular filling with sodium chloride 0.9% (10mL/kg during 10 min).
* Written, informed consent obtained from the 2 parents

Exclusion Criteria:

* Allergy to Ephedrine.
* Emergency surgery.
* Patient having previously received other vasopressive amines.
* Use of other indirect sympathomimetic drug such as phenylpropanolamine, phenylephrine, pseudoephedrine and methylphenidate.
* Premedication with clonidine
* Congenital heart disease
* IV-induced anesthesia.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
Therapeutic success is defined as a mBP superior to 55% of the basal mBP (prior to anesthesia) within 10 minutes post Ephedrine administration | Continuous monitoring within 10 minutes post-administration

SECONDARY OUTCOMES:
Return to a mBP superior to 38mmHg within 10 minutes post Ephedrine administration | Continuous monitoring within 10 minutes post-administration
Variations of O2 saturation in cerebral tissue (number of desaturations, evolution under treatment) using a Near Infrared Spectroscopy (NIRS) technology | Continuous monitoring within 10 minutes post-administration
Tolerance of Ephedrine: occurrence of serious adverse events | During 3 days post-administration
  Clinical examination focusing specifically on heart rate and hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde de Queiroz Siqueira, MD, Principal Investigator — Service d'anesthésie pédiatrique et obstétricale, Hôpital Femme Mère Enfant, 59 boulevard Pinel - 69 677 BRON Cedex
Locations (3):
- France (3):
  - Hôpital d'Estaing, Clermont-Ferrand
  - Hospices Civils de Lyon, Lyon
  - Hôpital Nord, Saint-Etienne

REFERENCES:
- [Result] Szostek AS, Saunier C, Elsensohn MH, Boucher P, Merquiol F, Gerst A, Portefaix A, Chassard D, De Queiroz Siqueira M. Effective dose of ephedrine for treatment of hypotension after induction of general anaesthesia in neonates and infants less than 6 months of age: a multicentre randomised, controlled, open label, dose escalation trial. Br J Anaesth. 2023 May;130(5):603-610. doi: 10.1016/j.bja.2022.12.006. Epub 2023 Jan 12. PMID 36639328
- [Derived] Szostek AS, Boucher P, Subtil F, Zerzaihi O, Saunier C, de Queiroz Siqueira M, Merquiol F, Martin P, Granier M, Gerst A, Lambert A, Storme T, Chassard D, Nony P, Kassai B, Gaillard S. Determination of the optimal dose of ephedrine in the treatment of arterial hypotension due to general anesthesia in neonates and infants below 6 months old: the ephedrine study protocol for a randomized, open-label, controlled, dose escalation trial. Trials. 2021 Mar 12;22(1):208. doi: 10.1186/s13063-021-05155-2. PMID 33712076